CLINICAL TRIAL: NCT04814355
Title: The Effect of Celecoxib on Neuroinflammation in MDD: PET Imaging of a Novel Treatment Target With [18F]FEPPA
Brief Title: The Effect of Celecoxib on Neuroinflammation in MDD
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Christine DeLorenzo, Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 81741
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder; Neuroinflammation
Keywords: PET; Major Depressive Disorder; Neuroinflammation
MeSH Terms: conditions — Depressive Disorder, Major; Neuroinflammatory Diseases | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Celecoxib 400 mg (Experimental): Patients will receive 400 mg/day of celecoxib for 8 weeks.
  Interventions: Drug: Celecoxib 400 mg

INTERVENTIONS:
Drug: Celecoxib 400 mg — Patients will receive 400 mg/day of celecoxib for 8 weeks.
  Other Names: celebrex

SUMMARY:
Major depressive disorder (MDD) affects an estimated 350 million people worldwide and is a leading contributor to global disease burden. Commonly used monoamine reuptake-inhibiting treatments for depression are suboptimal, resulting in only 30% of patients achieving remission. This may be because monoamine dysfunction is not the primary pathophysiology in all MDD patients. One avenue for the development of novel MDD treatments is through anti-inflammatory drugs; MDD is linked to a pro-inflammatory phenotype characterized by microglial activation, leading to the release of pro-inflammatory cytokines and upregulation of cellular markers including cyclooxygenase-2 (COX-2) and translocator protein (TSPO; a protein located on the outer membrane of microglia). Relevant to this proposal, TSPO can serve as an in vivo marker of neuroinflammation using the newly developed positron emission tomography (PET) tracer for TSPO, [18F]FEPPA. In support of this, a recent [18F]FEPPA PET study found that MDD patients in a current major depressive episode (MDE) had significantly higher TSPO binding in the prefrontal cortex (PFC), anterior cingulate cortex (ACC) and insula, relative to healthy controls. The prefrontal cortex and ACC are both implicated in mood regulation whereas the insula is involved in interoceptive signaling, which is known to be abnormal in MDD. Celecoxib, a selective COX-2 nonsteroidal anti-inflammatory drug (NSAID), is a promising new treatment for neuroinflammation in MDD. Clinical studies have observed that, in a subset of depressed patients, celecoxib treatment reduced depression severity as assessed by the Hamilton Depression Rating Scale (HDRS). While these findings demonstrate that celecoxib reduces symptom severity, PET imaging technology is critical for understanding how celecoxib affects the underlying pathophysiology of depression. Here, the team will investigate neuroinflammation as an underlying pathology in depression and test whether neuroinflammation is reduced by celecoxib in MDD patients. Specifically, in the proposed pilot study, MDD patients in a current MDE will receive [18F]FEPPA PET scans prior to and following 8 weeks of treatment with 400mg/day of celecoxib, with HDRS scores obtained at each time point. The investigators hypothesize that following celecoxib treatment, patients will show a significant reduction in neuroinflammation in the PFC, ACC and insula, which will correlate positively with the reduction in depressive symptoms, as measured by the HDRS. The proposed study will use novel imaging technology, [18F]FEPPA PET, to measure the effects of celecoxib on neuroinflammation in MDD patients. Our results will help to 1) identify neuroinflammation as an underlying pathology in MDD and 2) test whether reduction of inflammation is the mechanism of action of celecoxib. As such, the results of this study will aid in the development of targeted clinical treatments to improve remission rates in MDD patients.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-65
* Diagnosis of MDD and currently in a major depressive episode
* Capacity to give informed consent
* Score of at least 29 on the MADRS

Exclusion Criteria

* Low affinity binders (LABs) for TSPO Genotype
* Hypersensitivity to celecoxib, sulfonamides, aspirin, other NSAIDs, or any component of the formulation; previous asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs
* Heptic impairment, heart failure, severe renal impairment, recent GI bleed, history of peptic ulcer disease, anemia or any other contraindication for celecoxib
* Poor CYP2C9 metabolizer
* Currently taking medications that interact with celecoxib (digoxin, antihypertensives, diuretics, anticoagulant or anti-platelet treatment, including aspirin)
* Use of herbs, drugs, or medications with anti-inflammatory or immunomodulatory properties (within 5 half-lives of starting celecoxib treatment)
* Unlikely to tolerate medication washout or the medication-free period following washout
* Participant considered at significant risk for suicide
* ECT within 1 month
* High potential for excessive drug/alcohol use during the treatment period (excluding nicotine or cannabis)
* Significant active physical illness or neurological deficit that may affect brain functioning or imaging
* Any PET contraindications, including if study imaging will result in the participant receiving greater exposure than the research limit, or if participant is currently pregnant, breastfeeding, or planning to conceive during the course of study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in neuroinflammation as measured by [18F]FEPPA PET. | Before and after 8 weeks of treatment with celecoxib.
  Change in [18F]FEPPA VT (VT; volume of distribution: ratio of the concentration of radioligand in tissue to that in plasma at equilibrium)

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 (HAMD) score. | Before and after 8 weeks of treatment with celecoxib.
  Comparison of Hamilton Depression Rating Scale-17 score at pretreatment and post-treatment. Minimum score 0, maximum possible score 52, with remission defined as <=7. The higher the score on the scale, the more severe the degree of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Christine DeLorenzo, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Psychiatry Department at Stony Brook University, Stony Brook, New York, United States